CLINICAL TRIAL: NCT00709800
Title: A Phase 1, Double-Blinded Study to Evaluate the Safety, Tolerability, and Immunogenicity of Pandemic Influenza Plasmid DNA Vaccines
Brief Title: Pandemic Influenza Plasmid DNA Vaccines (Needle)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vical (Industry)
Responsible Party: Don Guterwill, BS, MT, Senior Clinical Project Manager, Vical Incorporated
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: IPT1-101
Record Dates: First submitted 2008-07-01; First posted 2008-07-03 (Estimated); Last update posted 2009-02-12 (Estimated); Status verified 2009-02

CONDITIONS: Influenza
Keywords: Pandemic Influenza; Avian Influenza; DNA Vaccines; Antibody; T Cells; HA/NP/M2
MeSH Terms: conditions — Influenza, Human; Influenza in Birds

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- 2 (Experimental)
  Interventions: Biological: VCL-IPT1
- 3 (Experimental)
  Interventions: Biological: VCL-IPT1
- 4 (Experimental)
  Interventions: Biological: VCL-IPM1
- 5 (Placebo Comparator)
  Interventions: Biological: PBS
- 1 (Experimental)
  Interventions: Biological: VCL-IPT1

INTERVENTIONS:
Biological: VCL-IPT1 — IM, 0.1 mg/mL, 2 injections, 0 and 21 days
  Arms: 1
Biological: VCL-IPT1 — IM, 0.5 mg/mL, 2 injections, 0 and 21 days
  Arms: 2
Biological: VCL-IPT1 — IM, 1 mg/mL, 2 injections, 0 and 21 days
  Arms: 3
Biological: VCL-IPM1 — IM, 1 mg/mL, 2 injections, 0 and 21 days
  Arms: 4
Biological: PBS — IM, 1 mL, 2 injections, 0 and 21 days
  Other Names: Phosphate Buffered Saline
  Arms: 5

SUMMARY:
The trial will enroll up to 57 subjects. Qualified normal healthy volunteers will be enrolled in the study to receive the vaccine or placebo vaccine. Subjects will receive 2 vaccinations with a needle and will be followed for 6 months to evaluate the safety of and the immune system's response to the vaccine. The safety and immune system response will be studied throughout the trial.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 45 years of age
* Able to provide informed consent and be followed for 6 months

Exclusion Criteria:

* No immunomodulatory therapy within the past 6 months
* No evidence of immunodeficiency or pregnancy
* No laboratory or evidence of clinically significant medical disease
* No history of previous pDNA immunization
* No influenza immunization within the past 30 days
* No blood donations within 30 days of screening visit
* No history of bleeding disorder
* No use of aspirin and/or anticoagulants within 2 weeks of the administration of the investigational vaccines

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2007-08; Primary Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Safety and Tolerability of VCL-IPT1 and VCL-IPM1 in adult subjects | 6 months

SECONDARY OUTCOMES:
Influenza-specific immunogenicity of VCL-IPT1 and VCL-IPM1 | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Don Guterwill, BS, MT, Study Chair — Vical
Locations (3):
- United States (3):
  - Accelovance, San Diego, California
  - SNBL, Baltimore, Maryland
  - SUNY at Stonybrook, Stony Brook Medical Center, Stony Brook, New York